CLINICAL TRIAL: NCT01055704
Title: Effect of Methylnaltrexone on Gastrointestinal and Colonic Transit in Health
Brief Title: Effect of Methylnaltrexone on GI Transit in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Michael Camilleri, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-002996
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2011-08-08 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Gastric Motility Disorder
Keywords: Methylnaltrexone; Codeine; Gastrointestinal motility; Colonic transit
MeSH Terms: interventions — methylnaltrexone; Codeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Methylnaltrexone (Experimental)
  Interventions: Drug: Methylnaltrexone only
- Codeine (Experimental)
  Interventions: Drug: Codeine only
- Methylnaltrexone + codeine (Experimental)
  Interventions: Drug: Methylnaltrexone + codeine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo + placebo

INTERVENTIONS:
Drug: Methylnaltrexone only — 0.30 mg/kg subcutaneous injection daily
  Other Names: MNTX; Relistor
  Arms: Methylnaltrexone
Drug: Codeine only — 30 mg taken orally four times daily for 5 days
  Arms: Codeine
Drug: Methylnaltrexone + codeine — Methylnaltrexone 0.30 mg/kg by subcutaneous injection once daily and codeine 30 mg taken orally four times daily for 5 days
  Arms: Methylnaltrexone + codeine
Drug: Placebo + placebo — Placebo subcutaneous injection once daily and placebo taken orally four times daily for 5 days
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double blind, placebo-controlled study evaluating the effects of placebo, codeine, methylnaltrexone and codeine with methylnaltrexone on gastrointestinal motility and colonic transit of solids in healthy human subjects.

The hypotheses are:

1. Methylnaltrexone administered subcutaneously enhances gastrointestinal motility with acceleration of overall colonic transit, and ascending colon emptying of solids in healthy humans.
2. Methylnaltrexone significantly accelerates colonic transit that is delayed by codeine

DETAILED DESCRIPTION:
Methodology

Following the initial screening visit (visit 1), participants will be randomized to study medication, either 0.30mg/kg methylnaltrexone subcutaneously or placebo once daily and 30 mg codeine orally or placebo taken four times daily for a total of five days. Participants will be randomly assigned to study medication and allocation will be concealed. A urine pregnancy test will be performed for all females of child bearing potential within the 48 hours prior to the receipt of study medication. Note that females who are status post bilateral tubal ligation, hysterectomy or postmenopausal are exempted from this test. Study medication will be administered on study med days 1, 2 and 3 (visits 2, 3 and 4) at the Clinical Research Unit (CRU). Participants will return for scintigraphic assessment of gastric, small bowel and colonic transit of solids on study med days 4 and 5 (visits 5 and 6). The transit studies will be undertaken on over a 48 hour time period; no study medication is given on the final day of transit (visit 7).

Investigational product, dosage, mode of administration, duration of treatment

0.30 mg/kg methylnaltrexone or placebo subcutaneously once daily and 30 mg codeine or placebo orally four times daily for five consecutive days.

Treatment groups

1. placebo + placebo (8 participants)
2. placebo + codeine 120mg (8 participants)
3. methylnaltrexone 0.30 mg/kg + placebo (16 participants)
4. methylnaltrexone 0.30 mg/kg + codeine 120 mg (16 participants)

Efficacy assessments

1. Scintigraphic gastrointestinal and colonic transit
2. Assessment of bowel pattern frequency and consistency made by the patient using the bowel pattern diary

Safety assessments

No safety assessments (routine laboratory analysis, ECG etc) will be performed as both methylnaltrexone and codeine are FDA approved medications

Statistical analysis

The overall effects of the methylnaltrexone treatment on the primary and secondary response measures will be assessed using an analysis of covariance (ANCOVA) with suitable transformation for skewness in the distributions of measured responses if necessary (e.g., ANCOVA on ranks or an arcsine square root transformation for the proportion of marker in the colon at 6 hours). The covariates considered for inclusion in the analyses will be age, gender and body mass index. An a priori anticipated contrast (overall drug vs. placebo) will be examined (α = 0.05). The specific comparisons of methylnaltrexone vs placebo and codeine vs codeine plus methylnaltrexone are of significant interest, and since they are related to specific hypotheses, no change in α from 0.05 is planned.

ELIGIBILITY:
Inclusion Criteria

* Males and non-pregnant, non-breastfeeding females
* 18-65 years old
* No functional GI disorders on the short Bowel Disease Questionnaire (BDQ)
* A BMI greater than 22.0

Exclusion criteria

* Structural or metabolic diseases/conditions that affect the gastrointestinal system or functional gastrointestinal disorders. The short version of the Bowel Disease Questionnaire (BDQ) will be exclude functional GI disorders. More than three positive responses will exclude participation.
* Unable to withdraw from the following medications 48 hours prior to study entry:Any medication that alters GI transit including but not limited to laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, SSRI and newer antidepressants; analgesic drugs including opiates, NSAID, COX 2 inhibitors (note : Tylenol is permitted); GABAergic agents and benzodiazepines. Note: Concomitant medications will be reviewed on a case by case basis by the study physicians.
* Subjects who are considered by the investigator to be alcoholics not in remission or known substance abusers. Alcohol must be avoided from seven days prior to beginning the study medication until the completion of the study.
* Subjects who have participated in another clinical study within the past 30 days.
* Clinical evidence (including physical exam and review of the medical history) of significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Wong BS, Rao AS, Camilleri M, Manabe N, McKinzie S, Busciglio I, Burton DD, Ryks M, Zinsmeister AR. The effects of methylnaltrexone alone and in combination with acutely administered codeine on gastrointestinal and colonic transit in health. Aliment Pharmacol Ther. 2010 Oct;32(7):884-93. doi: 10.1111/j.1365-2036.2010.04422.x. PMID 20839388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants included males and non-pregnant, non-breastfeeding females aged 18 to 55 years. All subjects had a minimum body mass index (BMI) of 22 kg/m2.
Pre-assignment Details: Subjects were screened for eligibility within 28 days of Day 1 of the study. They were stratified based on gender and BMI (<25, ≥25 kg/m2) and randomized into one of four treatment groups: Treatment groups were randomly assigned in fixed block sizes according to a schedule provided by the study statistician (ARZ). Allocation sequence was concealed
Period: Overall Study
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Started | 16 | 8 | 16 | 8
Completed | 16 | 8 | 16 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 16 | 8 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 8 | 16 | 8 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.9 (2.6) | 39.4 (3.8) | 31.6 (2.7) | 36.1 (3.6) | 37.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 10 | 5 | 31
  Male | 5 | 3 | 6 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Colonic Geometric Center at 24 Hours
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit. A GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Units on a scale | 2.3 (0.2) | 1.8 (0.2) | 1.9 (0.3) | 2.3 (0.4)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.902, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -0.048, 95% CI 2-sided [-0.835 to 0.739], Standard Error of Mean 0.389
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.709, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = 0.132, 95% CI 2-sided [-0.578 to 0.841], Standard Error of Mean 0.351

2. Secondary Outcome: T1/2 of Ascending Colon Emptying
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: hours
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
hours | 17.1 (2.2) | 24.0 (3.9) | 23.6 (3.3) | 14.1 (2.6)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.675, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -1.971, 95% CI 2-sided [-11.415 to 7.472], Standard Error of Mean 4.669
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.591, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -2.280, 95% CI 2-sided [-10.792 to 6.233], Standard Error of Mean 4.208

3. Secondary Outcome: T1/2 of Gastric Emptying of Solid
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Minutes | 102.7 (5.1) | 104.0 (14.1) | 126.8 (11.9) | 101.1 (6.2)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.024, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Median Difference (Final Values) = -34.425, 95% CI 2-sided [-64.097 to -4.753], Standard Error of Mean 14.670
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.989, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Median Difference (Final Values) = -0.181, 95% CI 2-sided [-26.962 to 26.598], Standard Error of Mean 13.240

4. Secondary Outcome: Colonic Geometric Center at 4 Hours
Description: as for outcome 1
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Units on a scale | 0.236 (0.105) | 0 (0) | 0.379 (0.130) | 0.347 (0.229)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.064, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -0.401, 95% CI 2-sided [-0.827 to 0.025], Standard Error of Mean 0.211
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.610, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [-0.287 to 0.482], Standard Error of Mean 0.190

5. Secondary Outcome: Colonic Geometric Center at 48 Hours
Description: as for outcome 1
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Units on a scale | 3.9 (0.3) | 3.3 (0.4) | 2.8 (0.3) | 4.1 (0.2)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.151, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = 0.728, 95% CI 2-sided [-0.278 to 1.734], Standard Error of Mean 0.497
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.806, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [-0.795 to 1.017], Standard Error of Mean 0.448

6. Secondary Outcome: Colonic Filling at 6 Hours
Description: Percent of solids reaching the colon at 6 hours
Time Frame: 6 hours
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Percentage | 21.9 (5.7) | 23.7 (11.2) | 28.0 (6.9) | 34.5 (14.1)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI as covariates; Test type: Superiority or Other; p = 0.889, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = 1.772, 95% CI 2-sided [-23.678 to 27.223], Standard Error of Mean 12.583
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.274, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = 12.607, 95% CI 2-sided [-10.362 to 35.577], Standard Error of Mean 11.356

7. Secondary Outcome: Stool Frequency
Description: Stool frequency was self reported in a daily bowel pattern diary for 13 days.
Time Frame: daily
Measure: Mean (Standard Error); unit: Stools
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Stools | 1.1 (0.1) | 0.63 (0.2) | 0.7 (0.1) | 1.5 (0.4)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.236, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -0.214, 95% CI 2-sided [-0.572 to 0.145], Standard Error of Mean 0.178
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.885, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.412 to 0.357], Standard Error of Mean 0.190

8. Secondary Outcome: Stool Consistency as Reported From the Bristol Stool Scale
Description: Bristol Stool Scale a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation, with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
Time Frame: Daily
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Number analyzed (Participants) | 16 | 8 | 16 | 8
Units on a scale | 3.4 (0.3) | 3.1 (0.5) | 3.3 (0.3) | 3.7 (0.3)
Statistical Analysis 1: Comparison: Codeine 30 mg vs Methylnaltrexone 0.30 mg/kg + Codeine 30 mg; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.192, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -0.497, 95% CI 2-sided [-1.255 to 0.261], Standard Error of Mean 0.374
Statistical Analysis 2: Comparison: Methylnaltrexone 0.30 mg/kg vs Placebo; Data were analyzed using analysis of covariance (ANCOVA) with gender and/or BMI included as covariates; Test type: Superiority or Other; p = 0.855, ANCOVA; Error degrees of freedom adjusted for number of missing values imputed; Mean Difference (Final Values) = -0.063, 95% CI 2-sided [-0.756 to 0.630], Standard Error of Mean 0.342

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Methylnaltrexone 0.30 mg/kg | Codeine 30 mg | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 12/16 | 7/8 | 11/16 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylnaltrexone 0.30 mg/kg (N=16) | Codeine 30 mg (N=8) | Methylnaltrexone 0.30 mg/kg + Codeine 30 mg (N=16) | Placebo (N=8)
Burn or sting with injection (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) | 2 (2) | 5 (5)
Fatigue (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (2)
Headache (General disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Sleepiness (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Abdominal bloating (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
We did not evaluate dose-response. A higher dosage of MNTX may be needed to produce a detectable effect on GI and colonic transit as well as bowel pattern in healthy subjects who are naive to opioid agonists during MNTX initiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No